CLINICAL TRIAL: NCT02006784
Title: Pilot Study in Children With Systemic Lupus Erythematosus (SLE) to Assess Flares and to Measure Traditional and Novel Blood Biomarkers and Antibody Titers Following Receipt of Inactivated Influenza Vaccine (IIV)
Brief Title: Pilot Study to Assess Flares Following Inactivated Influenza Vaccine in Children With Systemic Lupus Erythematosus (SLE)
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Collaborators: Vanderbilt University Medical Center (Other); Baylor Research Institute (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kathryn Edwards, Professor of Pediatrics, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Other Study IDs: CISA 2013 TASK II
Record Dates: First submitted 2013-12-04; First posted 2013-12-10 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Systemic Lupus Erythematosus (SLE)
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum Blood
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an open label, pilot, observational, prospective study of the safety of inactivated influenza vaccine (IIV) in children with systemic lupus erythematosus (SLE) to be conducted during the 2013-2014 influenza season. The study will test conventional and novel biomarkers to assess disease flare and vaccine response and will also collect self-reported signs/symptoms in reactogenicity diaries during the 14 days after vaccination.

DETAILED DESCRIPTION:
This is an open label, pilot, observational, prospective study of the safety of inactivated influenza vaccine (IIV) in children with systemic lupus erythematosus (SLE) to be conducted during the 2013-2014 influenza season.

Annual receipt of IIV is recommended for persons with SLE and is considered a standard of care medical practice. The study will test conventional and novel biomarkers to assess disease flare and vaccine response and will also collect self-reported signs/symptoms in reactogenicity diaries during the 14 days after vaccination.

Little is known about the immune responses to influenza and other vaccines in children and adolescents with autoimmune conditions, both in terms of immunogenicity as well as the potential for triggering or worsening of immune/autoimmune pathways. Patients with SLE often must take two or more immunosuppressive medications to control their illness. Thus, it is critically important to study vaccine safety and immunogenicity within the pediatric SLE population rather than extrapolate the limited data available from adult clinical studies. Newly diagnosed, untreated patients will be too sick to include in this study. After that, patients are on some immunosuppressive regimen for an extended period of time.

This project will inform the process for a subsequent larger multi-center study to assess IIV safety utilizing an established clinical research network in pediatric rheumatology, such as the Childhood Arthritis and Rheumatology Research Alliance (CARRA) or other venue.

The pilot study will enroll 30 children with mild to moderate SLE as defined by a Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) of <6. A SLEDAI score is an SLE Disease Activity Index which consists of 24 items made up of both clinical data and laboratory results. This score is assessed each time that a patient with SLE is seen in the clinic. It is anticipated that the subjects would be enrolled over 2 to 3 months prior to the influenza season, so as to immunize the SLE patients with IIV before they would be exposed to the circulating wild-type influenza virus. Patients will be followed for 3 months.

Thirty patients receiving one of two different treatment regimens that are standard-of-care regimes, "Prednisone + Hydroxychloroquine" or Prednisone+ Hydroxychloroquine + Mycophenolate Mofetil (MMF), will be observed. All subjects will receive US-licensed influenza vaccines as part of standard medical practice.

These two regimens were chosen because they represent customary care immunosuppressant medication regimens for persons with SLE. In addition, MMF in the second treatment arm has an inhibitory effect on plasma cell development, therefore allowing us to explore whether patients receiving this drug will have diminished antibody responses in response to vaccination.

Fifteen patients will already be receiving Prednisone + Hydroxychloroquine and 15 patients will already be receiving Prednisone+ Hydroxychloroquine + Mycophenolate Mofetil (MMF) as their routine care

ELIGIBILITY:
Inclusion Criteria:

INCLUSION CRITERIA:

Subjects who meet the following criteria will be allowed to participate in the study:

1. Complete immunization history must be available at time of enrollment
2. Patients will be aged 8-18 years at time of enrollment
3. Patient will have stable disease activity (no changes in SLEDAI >2 points) during the 3 months preceding enrollment.
4. Patients can be enrolled as soon as the seasonal IIV is available and prior to the onset of influenza activity in the community. Generally this will be between September 2013-January2014. If feasible, enrollment will end in December 2013, which is usually before influenza circulates widely in the community.

Exclusion Criteria:

Subjects who meet the following criteria will not be allowed to participate in the study:

1. Females who are known to be pregnant or breastfeeding
2. Moderate to high SLE disease activity at enrollment (SLEDAI >6)
3. Oral temp ≥100F (≥37.8) within 72 hours prior to vaccination
4. History of allergy to egg or egg products or history of allergic reaction to previous influenza vaccination or vaccine constituent
5. History of Guillain-Barré syndrome after previous immunizations
6. Unstable SLE disease activity during 3 months prior to enrollment (change in SLEDAI score >2)
7. Requirement for high-dose IV Solumedrol and/or Cytoxan pulse therapy during 6 months prior to study
8. Any condition that study site investigator deems would put patient at unacceptable risk of injury or render patient unable to meet requirements of the protocol.
9. Received pre-medication with analgesic or antipyretic agents in the 6 hours prior to first vaccination, or planned medication with analgesic or antipyretic in the week following first vaccination. This criterion should not preclude subjects receiving such medication if the need arises. However, pre-medication is to be discouraged.
10. Patient has received other inactivated vaccines within 14 days prior to administration of IIV.
11. Patient is scheduled to receive another routinely administered inactivated vaccine within 14 days after IIV.
12. Patient is currently participating in a study that involves and experimental agent (vaccine, drug, biologic, device, blood product, or medication), or expects to receive another experimental agent during participation in this study

    -

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study will recruit and enroll thirty pediatric patients, 8-18 years of age,with a diagnosis of mild to moderate (SLEDAI < 6) Systemic Lupus Erythematosus, who are seen for routine clinic visits in the rheumatology clinics at Texas Scottish Rite Hospital and Children's Medical Center, Dallas, TX during the 2013-2014 influenza seasons. Treatment Arms 1 and 2 will be comprised of patients with similar demographics in terms of race, ethnicity, and gender.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
To assess the achievability of the pilot protocol | 18 months
  * Ability to recruit the entire sample cohort of 30 subjects during the pre-planned enrollment period.
  * Eighty percent of subjects complete all blood draws within the designated time frame
  * Adherence to protocol for blood collection, reaction assessment, clinic follow up, and laboratory analysis for 80% of the enrolled cohor

SECONDARY OUTCOMES:
Lupus Flares | 90 days
  * To ascertain the ability to detect flares and associate the flare to vaccine
  * To correlate post-vaccine changes in blood biomarkers with the development of flares as assessed by SLEDAI and BILAG scores as well as self- and physician-assessed reactogenicity
To assess immunogenicity of IIV in children with autoimmunity on two different immunosuppressive regimens | 90days
  * To ascertain the development of neutralizing and hemagglutination inhibition (HAI) antibody titers at baseline and at 28 days (+ 7 day)
  * To correlate changes in blood biomarkers with response to vaccine using immune profiling analysis.

CONTACTS AND LOCATIONS:
Overall Officials: M. Virginia Pascual, MD, Principal Investigator — Baylor Research Institute; Kathryn M Edwards, MD, Principal Investigator — Vanderbilt Medical Center; Theresa Harrington, MD, Principal Investigator — Centers for Disease Control and Prevention
Locations (1):
- Baylor Institute for Immunology Research, Dallas, Texas, United States